CLINICAL TRIAL: NCT01612130
Title: Valeriana Officinalis L. for Conscious Sedation in Patients Submitted to Impacted Lower Third Molars Surgery: A Randomized, Double-Blind, Placebo-Controlled Crossover Study
Brief Title: Valerian for Conscious Sedation in Patients Submitted to Impacted Lower Third Molars Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of the Valleys of Jequitinhonha and Mucuri (Other)
Collaborators: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Marcos Luciano Pimenta Pinheiro, Professor of Pharmacology and Therapeutics, Department of Basic Science, Biologic and Health Sciences Faculty, Federal University of Vales do Jequitinhonha e Mucuri - UFVJM, Diamantina, Minas Gerais, Brazil., Federal University of the Valleys of Jequitinhonha and Mucuri
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 098/2002
Record Dates: First submitted 2012-06-01; First posted 2012-06-05 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Dental Anxiety; Blood Pressure; Heart Rate
MeSH Terms: interventions — Valeriana extract

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Valeriana officinalis L (100mg) (Experimental): 100 mg of Valeriana officinalis L. (Valerian)
  Interventions: Drug: 100 mg of Valeriana officinalis L
- Placebo (100 mg) (Placebo Comparator): Placebo 100mg
  Interventions: Drug: Placebo 100mg

INTERVENTIONS:
Drug: 100 mg of Valeriana officinalis L — A single dose of 100 mg of Valeriana officinalis L., 1 hour prior to surgical procedures
  Other Names: Valerian
  Arms: Valeriana officinalis L (100mg)
Drug: Placebo 100mg — A single dose of 100 mg of placebo orally, 1 hour prior to surgical procedures
  Arms: Placebo (100 mg)

SUMMARY:
The aim of the present study was to evaluate the efficacy of Valeriana officinalis L. 100 mg in single oral doses one hour preoperative as conscious sedation during the impacted lower third molar surgery.

DETAILED DESCRIPTION:
Evaluate the efficacy of Valeriana officinalis L. (Valerian) for control of anxiety during third molar surgery. Study design: A single oral dose of either valerian (100 mg) or placebo was randomly administered one hour before each surgical procedure to 20 volunteers between 17 and 31 years of age. Anxiety level was assessed through questionnaires, physiological parameters (blood pressure and heart rate) and the observation of signs.

ELIGIBILITY:
Inclusion Criteria:

* Indication for bilateral extraction of asymptomatic impacted mandibular third molars in similar positions based on the Pell & Gregory classification

Exclusion Criteria:

* Use of any type of medication in the 15 days prior to the onset of the study; history of hypersensitivity to the drugs, substances or materials employed in the experiment; pregnancy or lactation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-03; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Signs and symptoms of anxiety | 1 day (during dental appointment)
  During each surgery, the researcher and surgeon observed the manifestation of signs and symptoms associated to anxiety (restlessness/agitation/nervous ticks, paleness, excessive perspiration, tingling sensation in hands, feet or lips, change in breathing rhythm or depth). In the presence of one or more of these signs and symptoms, the patient was classified as anxious. If there was no manifestation of anxiety, the patient was classified as calm or relaxed
assessment of the blood pressure | 1 day (during dental appointment)
  The assessment of the blood pressure was performed at three moments: baseline, post-medication and end of surgery.
Assesment of heart rate | 1 day (during dental appointment)
  The assessment of the heart rate was performed at three moments: baseline, post-medication and end of surgery.

SECONDARY OUTCOMES:
Oxygen saturation | 1 day (During dental appointment)
  Level of blood oxygen saturation 30 minutes after drug administration and throughout the surgical procedure.
Side effects of drugs | 1 week
  Evaluation of the incidence of side effects of drugs used were informed by the patient after de drug administration until one week of postoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Marcos Pinheiro, PhD, Principal Investigator — Federal University of the Valleys of Jequitinhonha and Mucuri
Locations (1):
- Oral-Maxillofacial Surgery Sector of the Piracicaba Dental School, Universidade Estadual de Campinas (Brazil), Piracicaba, São Paulo, Brazil